CLINICAL TRIAL: NCT00376753
Title: The Effect of Surround Inhibition During Phasic Compared to Tonic Voluntary Finger Movement in Focal Hand Dystonia
Brief Title: Muscle Contraction in Patients With Focal Hand Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060242; 06-N-0242
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-11

CONDITIONS: Focal Hand Dystonia
Keywords: Transcranial Magnetic Stimulation (TMS); Writer's Cramp; Electromyogram; Focal Hand Dystonia; FHD; Healthy Volunteer; HV
MeSH Terms: conditions — Dystonia, Focal, Task-Specific; Dystonic Disorders

SUMMARY:
This study will examine and compare brain activity in people with focal hand dystonia (FHD) and healthy volunteers to obtain further knowledge about the underlying cause of FHD. Patients with dystonia have muscle spasms that cause abnormal postures while trying to perform a movement; FHD affects the hands and fine finger movements. During fine finger movement, the brain controls muscles in a process called surround inhibition. This process may be impaired in people with hand dystonia, leading to uncontrolled overactivity in muscles and impairing motor function.

Healthy volunteers and patients with FHD over 18 years of age may be eligible for this study. Candidates are screened with a physical and neurological examination.

In a series of three experiments conducted during a single clinic visit, participants undergo transcranial magnetic stimulation (TMS) while performing a finger movement. A wire coil is placed on the subject's scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that travels through the scalp and skull and causes small electrical currents in the outer part of the brain. The stimulation may cause muscle, hand or arm twitching, or may affect movement or reflexes. During the stimulation, the subject is asked to contract one finger.

In addition to TMS, subjects have surface electromyography. For this test, they sit in a chair with their hands placed on a pillow on their lap. The electrical activity of three muscles in the right hand is recorded by electrodes (small metal disks) taped to the skin over the muscles.

DETAILED DESCRIPTION:
OBJECTIVE:

In sensory systems, a neural mechanism called surround inhibition (SI) sharpens sensation by creating an inhibitory zone around the central core of activation. This principle was described for the visual system first, but there is evidence for similar mechanisms in the primary motor cortex (M1) involved in movement generation and control, especially in precise motor tasks. Dystonia is generally regarded as a motor execution abnormality due to a dysfunction in the cortico-striato-thalamo-cortical motor loop. Using transcranial magnetic stimulation (TMS), recent findings point to highly task-specific impairment of motor cortical inhibition in patients with focal hand dystonia (FHD).

The goal for this research proposal is to understand the underlying physiology as it relates to different inhibitory pathways on movement generation and control. To achieve this goal, different modes of voluntary contractions will be examined in healthy controls and patients with FHD with the prospect of having new options for treatment.

STUDY POPULATION:

We intend to study 100 adult patients with FHD and 100 healthy volunteers on an outpatient basis.

DESIGN:

Participants will perform a contraction of the first dorsal interosseous muscle (FDI). At rest, before EMG-onset (premotor), during phasic and tonic contraction single TMS pulses (Experiment 1) or double TMS pulses (Experiment 2) will be applied over the primary motor cortex to assess activation-induced changes in cortical excitability in the abductor pollicis brevis muscle (APB), which is not activated. Additionally the influence of visual feedback on short intracortical inhibition (SICI) will be tested in Experiment 3. In Experiment 4-8 interhemispheric (IHI), ventral and dorso-lateral premotor-motor intracortical inhibition will be assessed.

OUTCOME MEASURES:

The primary outcome measure for Experiment 1 will be the difference in MEP peak-to-peak amplitude between all motor conditions.

The primary outcome measure for Experiment 2, 5, 6, 7 and 8 will be the difference in normalized MEP peak-to-peak amplitude between all motor conditions in FHD patients and healthy volunteers.

In Experiments 1 and 2, the change in MEP peak-to-peak amplitude between different force levels (10% versus 20%) will be a second outcome parameter.

The primary outcome parameter for Experiment 3 will be change in MEP peak-to-peak between patients and healthy volunteers during tonic contraction with and without visual feedback.

In Experiment 4, Hmax/Mmax ratio will be the primary outcome parameter.

ELIGIBILITY:
* INCLUSION CRITERIA:

PATIENTS:

18 years old or older

Presence of FHD, for Experiment 5, 6, 7 and 8 the affected limb has to be the right and dominant side

HEALTHY VOLUNTEERS:

18 years old or older

Right handedness

Absence of dystonia or other neurological disorder with any effect on the motor or sensory systems

EXCLUSION CRITERIA:

PATIENTS AND HEALTHY VOLUNTEERS:

Concurrent significant medical, surgical, neurological or psychiatric condition

Taking the following medications: antidepressants, anxiolytics, anticonvulsants, antipsychotics, antiparkinson, hypnotics, stimulants, and/or antihistamines

Patients- Received botulinum toxin injection within 3 months of starting the protocol

For TMS: Presence of pacemaker, implanted medical pump, metal plate or metal object in skull or eye

History of seizure disorder

Known history of hearing loss

For MRI: Presence of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, or shrapnel fragments. Welders and metal workers are also at risk for injury because of possible small metal fragments in the eye of which they may be unaware.

Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-09-11; Study Completion 2011-05-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Berardelli A, Rothwell JC, Hallett M, Thompson PD, Manfredi M, Marsden CD. The pathophysiology of primary dystonia. Brain. 1998 Jul;121 ( Pt 7):1195-212. doi: 10.1093/brain/121.7.1195. PMID 9679773
- [Background] Bressman SB, de Leon D, Raymond D, Greene PE, Brin MF, Fahn S, Ozelius LJ, Breakefield XO, Kramer PL, Risch NJ. The role of the DYT1 gene in secondary dystonia. Adv Neurol. 1998;78:107-15. No abstract available. PMID 9750907
- [Background] Defazio G, Aniello MS, Masi G, Lucchese V, De Candia D, Martino D. Frequency of familial aggregation in primary adult-onset cranial cervical dystonia. Neurol Sci. 2003 Oct;24(3):168-9. doi: 10.1007/s10072-003-0113-3. PMID 14598070